CLINICAL TRIAL: NCT01018940
Title: Influence of the Proton Pump Inhibitor Omeprazole on the Anti-Platelet of P2Y12 Antagonists in Subjects With Coronary and Peripheral Artery Disease
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 14882
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease; Peripheral Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens for platelet activity and genotyping
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Plavix
- Prasugrel

SUMMARY:
To determine if prasugrel is superior to clopidogrel in providing adequate antiplatelet effect in a high risk population that requires concomitant use of a Proton Pump Inhibitor (PPI).

DETAILED DESCRIPTION:
To evaluate if simultaneous treatment with the PPI omeprazole and a P2Y12 receptor antagonist will influence the effect of either clopidogrel and/or prasugrel on platelet reactivity in patients with Coronary Artery Disease (CAD) or Peripheral Arterial Disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 75 years of age
* Known or documented history of CAD or PAD prior to enrollment (a diagnosis of CAD may be based upon a positive stress test, prior documented acute coronary event, or angiographic demonstration of CAD; a diagnosis of PAD may be based upon an ankle-brachial index less than 0.9, or angiographic demonstration of PAD)
* Have not had thienopyridine therapy for at least 15 days before the study
* Have not had treatment with a PPI for at least 15 days before the study
* Are taking aspirin (75 to 325 mg/day) for at least one week prior to randomization

Exclusion Criteria:

* Have New York Heart association (NYHA) Class III and IV congestive heart failure
* Have any form of coronary revascularization (PCI or coronary artery bypass grafting [CABG]) planned to occur during the study
* Have undergone PCI or CABG within 30 days of entry to the study
* Have received a drug eluting endovascular stents in the past year
* Have any of the following:

  1. Prior history of hemorrhagic stroke or transient ischemic attack (TIA)
  2. Intracranial neoplasm, arteriovenous malformation, or aneurysm
  3. A body weight less than 60 kg
* Have prior history of GI ulcer disease or bleeding
* Have symptoms of dyspepsia or gastroesophageal reflux disease
* Have active internal bleeding or history of bleeding diathesis
* Have clinical findings, in the judgment of the investigator, associated with an increased risk of bleeding
* Have an International Normalized Ratio (INR) known to be >1.5 at the time of evaluation
* Have a platelet count of <100,000/mm3 at the time of screening, if known
* Have anemia (hemoglobin [Hgb] <10 gm/dL) at the time of screening, if known
* Are receiving or will receive oral anticoagulation or other antiplatelet therapy (other than aspirin) that cannot be safely discontinued for the duration of the study
* Are receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) that cannot be discontinued or require daily treatment with NSAIDs during the study.
* Are receiving corticosteroid therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Coronary or Peripheral Artery Disease
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Saucedo, MD, Principal Investigator — Dept of Cardiology
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States